CLINICAL TRIAL: NCT04610775
Title: The Cuff Size Blood Pressure Measurement Trial
Brief Title: Cuff(SZ): The Cuff Size Blood Pressure Measurement Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Vital Strategies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: IRB00252142
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-03

CONDITIONS: Hypertension; Blood Pressure; Cardiovascular Diseases; Cardiovascular Risk Factor
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (24):
- Small Cuff (0, +1, +2, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Small, Regular, Large, Small
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Small Cuff (0, +2, +1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Small, Large, Regular, Small
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Small Cuff ( +1, 0, +2, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Regular, Small, Large, Small
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Small Cuff ( +1, +2, 0, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Regular, Large, Small, Small
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Small Cuff ( +2, 0, +1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Large, Small, Regular, Small
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Small Cuff ( +2, +1, 0, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Large, Regular, Small, Small
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Regular Cuff (0, -1, +1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Regular, Small, Large, Regular
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Regular Cuff (0, +1, -1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Regular, Large, Small, Regular
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Regular Cuff (-1, 0, +1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Small, Regular, Large, Regular
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Regular Cuff (-1, +1, 0, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Small, Large, Regular, Regular
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Regular Cuff (+1, -1, 0, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Large, Small, Regular, Regular
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Regular Cuff (+1, 0, -1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Large, Regular, Small, Regular
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Large Cuff (-1, 0, +1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Regular, Large, Extra Large, Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Large Cuff (-1, +1, 0, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Regular, Extra Large, Large, Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Large Cuff (0, +1, -1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Large, Extra Large, Regular, Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Large Cuff (0, -1, +1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Large, Regular, Extra Large, Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Large Cuff (+1, 0, -1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Extra Large, Large, Regular, Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Large Cuff (+1, -1, 0, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Extra Large, Regular, Large, Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Extra Large Cuff (0, -2, -1, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Extra Large, Regular, Large, Extra Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Extra Large Cuff (0, -1, -2, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Extra Large, Large, Regular, Extra Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Extra Large Cuff (-1, 0, -2, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Large, Extra Large, Regular, Extra Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Extra Large Cuff (-1, -2, 0, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Large, Regular, Extra Large, Extra Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Extra Large Cuff (-2, -1, 0, 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Regular, Large, Extra Large, Extra Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements
- Extra Large Cuff (-2, 0, -1 0) (Other): The order of blood pressure cuffs used for participants randomized to this arm will be: Regular, Extra Large, Large, Extra Large
  Interventions: Other: Order of cuff sizes during blood pressure measurements

INTERVENTIONS:
Other: Order of cuff sizes during blood pressure measurements — Each participant will have 4 sets of 3 blood pressure measurements taken. The participants will be randomized to the order in which the cuff sizes are used.

SUMMARY:
To determine the impact of overcuffing (using a too-large cuff) and undercuffing (using a too-small cuff) on initial BP and average BP measurements when using an automated BP device, overall and stratified by appropriate cuff size

To determine if the impact over- or under-cuffing differs based on the following patient characteristics:

1. Hypertensive (≥140/90 based on triplicate measures using appropriately sized cuff) vs. non-hypertensive.
2. Arm circumference (continuous)
3. Obesity status

DETAILED DESCRIPTION:
The investigators propose a cross-sectional study of adult participants recruited from the community. Enrolled participants will have 2-3 sets of three automated BPs measured, each set with a different cuff size. To accomplish this, the investigators will utilize a 2-3 period cross-over design:

• Two or three different periods with 3 automated BP measurements, using a BP cuff that is:

* Appropriately sized based on mid-upper arm circumference ( standard)
* Too small (one size lower than appropriate)
* Too large (one size higher than appropriate)

Individuals in whom the smallest available cuff (small adult) and largest available cuff (extra-large cuff) is appropriate for their arm circumference will only be able to undergo two periods of BP measurements.

ELIGIBILITY:
Inclusion Criteria:

* 18-80

Exclusion Criteria:

* Presence of the following on both arms: rashes, gauze dressings, casts, edema, paralysis, tubes, open sores or wounds, withered arms, A-V shunts, or if blood has been drawn from arm within last week.
* Being mentally impaired, pregnant.
* Arm circumference exceeding 50 cm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Difference in systolic BP in appropriately-sized cuff vs. too small cuff | Up to 90 minutes
  Difference between (1) 1st systolic BP and (2) average of 3 systolic BP from measurements (mmHg).
Difference in systolic BP in appropriately-sized cuff vs. too large cuff | Up to 90 minutes
  Difference between (1) 1st systolic BP and (2) average of 3 systolic BP from measurements (mmHg).
Difference in diastolic BP in appropriately-sized cuff vs. too small cuff | Up to 90 minutes
  Difference between (1) 1st diastolic BP and (2) average of 3 diastolic BP from measurements (mmHg).
Difference in diastolic BP in appropriately-sized cuff vs. too large cuff | Up to 90 minutes
  Difference between (1) 1st diastolic BP and (2) average of 3 diastolic BP from measurements (mmHg).

SECONDARY OUTCOMES:
Difference in blood pressure based on hypertension status | Up to 90 minutes
  To determine the blood pressure difference based on hypertensive (≥140/90 based on triplicate measures using appropriately sized cuff) vs. non-hypertensive participants.
Difference in blood pressure based on arm circumference | Up to 90 minutes
  To determine the blood pressure difference based on arm circumference (continuous).
Difference in blood pressure based on BMI | Up to 90 minutes
  To determine the blood pressure difference based on normal BMI (<25 kg/m2) vs. overweight BMI (25 kg/m2-29.99 kg/m2) vs. Class I Obesity (30 kg/m2-34.99 kg/m2) vs. ≥Class II Obesity (>35 kg/m2).

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Brady, MD,Phd, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins ProHealth Research Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ishigami J, Charleston J, Miller ER 3rd, Matsushita K, Appel LJ, Brady TM. Effects of Cuff Size on the Accuracy of Blood Pressure Readings: The Cuff(SZ) Randomized Crossover Trial. JAMA Intern Med. 2023 Oct 1;183(10):1061-1068. doi: 10.1001/jamainternmed.2023.3264. PMID 37548984